CLINICAL TRIAL: NCT01906567
Title: İs There a Relationship Between Severity of Preeclampsia and Maternal Heavy Metal Levels?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, Ayse Kirbas, Ayse Kirbas, MD, Zekai Tahir Burak Women's Health Research and Education Hospital
Other Study IDs: zekai tahir burak heavy metal
Record Dates: First submitted 2013-07-05; First posted 2013-07-24 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-07

CONDITIONS: Mild Pre-eclampsia; Severe Preeclampsia
Keywords: cadmium; lead; mercury; preeclampsia; pregnancy
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: None Retained — maternal whole blood maternal hair umbilical whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- severe preeclamptic women: Severe preeclampsia is defined as the presence of 1 of the following symptoms or signs in the presence of preeclampsia:
  • SBP of 160 mm Hg or higher or DBP of 110 mm Hg or higher on 2 occasions at least 6 hours apart
  • Proteinuria of more than 5 g in a 24-hour collection or more than 3+ on 2 random urine samples collected at least 4 hours apart
  • Pulmonary edema or cyanosis
  • Oliguria (< 400 mL in 24 h)
  • Persistent headaches
  • Epigastric pain and/or impaired liver function
  • Thrombocytopenia
  • Oligohydramnios, decreased fetal growth, or placental abruption
- mild preeclamptic women: Mild preeclampsia is defined as the presence of hypertension (BP ≥140/90 mm Hg) on 2 occasions, at least 6 hours apart, but without evidence of end-organ damage in the patient.
- Healthy Pregnant Women: healthy pregnant women at term who not developed any complication of pregnancy

SUMMARY:
The purpose of this study, to investigate whether severity of preeclampsia is associated with altered levels of heavy metals (Cd, Hg, arsenic and Pb) in maternal blood, fetal blood, and maternal hair.

DETAILED DESCRIPTION:
The unfavorable effects of heavy metals on human health is well known. The main threats to human health from heavy metals are associated with exposure to lead, cadmium, mercury and arsenic. They may be toxic at the levels previously thought to have no adverse effect on human.In utero environmental exposures can have long term consequences to health and development.İn spite of what is known about the neurotoxicity from exposure to heavy metals, the health effects from co-exposure to these chemicals and the biologically effective doses are not known exactly.

Preeclampsia is associated with increased maternal and infant mortality and morbidity. The exact etiology is not clear. Several evidences indicate that various environmental factors and elements may play a role in pre-eclampsia.

significant increase in Pb, cadmium (Cd), copper (Cu) and magnesium (Mg) and decrease in zinc (Zn) in amniotic fluid are associated with preeclampsia. Pb as this metal has well known adverse effects on renal system and blood pressures Effects of Pb on reproductive system have been studied intensively, e.g. other pregnancy outcome and pregnancy hypertension.

However, the relationship between the severity of pre-eclampsia and heavy metal levels have not been investigated.

The purpose of this study, to investigate whether severity of preeclampsia is associated with altered levels of heavy metals (Cd, Hg, arsenic and Pb) in maternal blood, fetal blood, and maternal hair.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of preeclampsia (diagnosed per ACOG criteria)

Exclusion Criteria:

known chronic disease multipl pregnancies

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women with preeclampsia
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2013-07; Primary Completion 2013-09 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
increased levels of heavy metals in preeclamptic women | 6 months
  mercury, cadmium and lead levels in maternal blood and hair

CONTACTS AND LOCATIONS:
Overall Officials: ayse kirbas, md, Principal Investigator — Zekai Tahir Burak Women's Health Research and Education Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Zekai Tahir Burak Maternity Teaching Hospital, Ankara, Ankara
  - Zekai Tahir Burak Education and Research Hospital, Ankara

REFERENCES:
- See also: Maternal Blood Lead Levels and the Risk of Pregnancy-Induced Hypertension: The EDEN Cohort Study — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2790505/
- See also: Environmental lead level and pregnancy-induced hypertension. — http://ncbi.nlm.nih.gov/